CLINICAL TRIAL: NCT06888245
Title: Evaluation of the Effectiveness of Menstruation Education Given to Secondary School Students With and Without Animation
Brief Title: Effectiveness of Menstruation Education to Secondary School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Assoc. Prof. Dr., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OrduA1
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Menstruation; Education; Student; Animation
Keywords: Menstruation; Student; Education; Animation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-animated Menstruation Education Group (Experimental): Non-animated menstruation education will be given to this arm.
  Interventions: Other: Non-animated Menstruation Education
- Animated Menstruation Education Group (Experimental): Animated menstruation education will be given to this arm.
  Interventions: Other: Animated Menstruation Education
- Control Group (No Intervention): Participants in the control group will not be subjected to any intervention during the research process.

INTERVENTIONS:
Other: Non-animated Menstruation Education — Providing menstruation education to female secondary school students with Powerpoint support without animation.
  Arms: Non-animated Menstruation Education Group
Other: Animated Menstruation Education — Providing menstruation education to female secondary school students with Powerpoint and animation support.
  Arms: Animated Menstruation Education Group

SUMMARY:
Supporting adolescents with education about the menstruation process is important in terms of managing the process physically and mentally healthy and gaining lifelong positive health behaviors. Various narrative techniques including visuals, slides and animations are utilized in menstruation education for adolescents. Within the scope of these narrative techniques, technological tools are frequently used for learning purposes in adolescence. In technology-supported education, training that includes visual materials such as animations and multimedia software is very important. Presentations supported by various visuals and texts can be effective in trainings on mentoring. Presentations can appeal to students' visual senses and attract their attention. Animation is one of the technology-based applications that are frequently used in the education of adolescents and support education. The presentation can be animated or non-animated.

DETAILED DESCRIPTION:
It is stated that girls experiencing the process without having information about menarche causes negative emotions such as fear, anxiety, sadness and crying. In addition, it is emphasized that girls have difficulties in managing the menstruation process and that they should be supported to manage this process in a healthy way.. In addition, it is stated that adolescents' school absenteeism increases, academic achievement decreases and school dropouts occur due to their inability to manage the menstrual process in the school environment. In this context, it is important to inform and support adolescents about the problems experienced during menstruation and coping techniques. It is reported that adolescents' early adoption of correct knowledge, attitudes and behaviors towards the menstruation process will positively affect physiological and psychological health, body image and healthy sexual identity formation.

Supporting adolescents with education about the menstruation process is important in terms of managing the process in a physically and mentally healthy way and gaining lifelong positive health behaviors. In mentoring education for adolescents, various visual, slide and animation narrative techniques are used. Within the scope of these expression techniques, technological tools are frequently used for learning purposes in adolescence. In technology-supported education, trainings that include visual materials such as animations and multimedia software are very important. Presentations supported by various visuals and texts can be effective in trainings on mentoring. Presentations can appeal to students' visual senses and attract their attention. Animation is one of the technology-based applications that are frequently used in the education of adolescents and support education. The presentation can be animated or non-animated. Animation is "the act of animating successive frames of connected movement within a period of seconds". It is stated that the use of animation in the education process concretizes complex subjects, increases retention, provides a fun learning experience, facilitates the learning of complex and difficult concepts, reinforces learning by emphasizing visuality, and is effective in drawing attention to the subject. In studies conducted on adolescent students, animation-supported education programs are reported to be more effective than presentation-supported lectures. In this context, it is important to provide animation-supported trainings to adolescents by health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Secondary school student
* Open to communication and collaboration,
* Female students who agreed to participate in the study and whose parents gave their consent were included in the study.

Exclusion Criteria:

* Special education students from the research,
* Female students who do not want to continue the research will be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Girls will be included in the study due to the evaluation of the effectiveness of menstruation education given within the scope of the study.
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge Test | From enrollment to the end of education at 2 weeks
  This knowledge test was developed by Gümüş (2024) to measure the knowledge level of middle school students about menstruation. In the knowledge test, "1 point" was given for a correct answer and "0 point" for an incorrect answer. The Kuder-Richardson (KR-20) value was found to be 0.563 to determine the internal consistency of the knowledge test.

IPD SHARING:
Plan to Share IPD: No